CLINICAL TRIAL: NCT00448812
Title: Extension Study for the Multicenter Randomized Clinical Trial of the Alair® System for the Bronchial Thermoplasty Treatment of Asthma (NCT00214526)
Brief Title: AIR Extension Study - Long-Term Safety of Alair Treated Subjects
Acronym: AIRx
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 05-01
Record Dates: First submitted 2007-03-16; First posted 2007-03-19 (Estimated); Results first posted 2021-02-17 (Actual); Last update posted 2021-02-17 (Actual); Status verified 2021-01

CONDITIONS: Asthma
Keywords: Alair System; Bronchial Thermoplasty; Long-term Safety
MeSH Terms: conditions — Asthma | interventions — Bronchial Thermoplasty

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Alair Treatment (Experimental): Subjects from PREDECESSOR STUDY (NCT00214526) treated with conventional therapy with ICS+LABA (inhaled corticosteroid + long-acting beta-agonist) plus Bronchial Thermoplasty with the Alair System.
  Interventions: Device: Bronchial Thermoplasty with the Alair System
- Control (No Intervention): Control group subjects from PREDECESSOR STUDY (NCT00214526).

INTERVENTIONS:
Device: Bronchial Thermoplasty with the Alair System — Treatment of airways with the Alair System (Bronchial Thermoplasty) in the PREDECESSOR STUDY (NCT00214526).
  Arms: Alair Treatment

SUMMARY:
The primary purpose of this study is to gather additional safety data for subjects who previously completed the one-year study entitled: "Multicenter Randomized Clinical Trial of the Alair System for the Bronchial Thermoplasty Treatment of Asthma" (Protocol #0602-20, NCT00214526) sponsored by Asthmatx, Inc. Study Subjects who were assigned to the Control Group who elect to participate in this extension study will be followed for an additional two (2) - year period beyond the PREDECESSOR STUDY'S one-year endpoint. Subjects treated with the Alair System who elect to participate in this extension study will be followed for an additional four (4)- year period beyond the PREDECESSOR STUDY'S one-year endpoint.

All treatments with the Alair System were completed in the PREDECESSOR STUDY (NCT00214526). The current study is designed solely to collect longer-term follow-up data on the effects of the treatments. The data will be of the same type that was collected in the PREDECESSOR STUDY (NCT00214526), including spirometry, physical examinations, review of symptoms, use of maintenance and rescue medications, and response to Methacholine challenge.

DETAILED DESCRIPTION:
This will be a multicenter study conducted only at the clinical sites that participated in the PREDECESSOR STUDY (NCT00214526).

Written, informed consent will be obtained prior to performing any study procedures. Enrollment will be limited to only those subjects who were in either the Control or Treatment groups of the PREDECESSOR STUDY (NCT00214526).

The present study will extend the follow-up evaluation of subjects from the PREDECESSOR STUDY (NCT00214526) to 3 years post-treatment for the Control Subjects and 5 years post-treatment for Alair-Treated Subjects. These evaluations will consist of two (Control Group) to four (Alair Group) additional study visits corresponding to the two-year, three-year, four-year and five-year time points following completion of Alair treatments (or similar time point for control subjects) in the PREDECESSOR STUDY (NCT00214526). For consistency with the PREDECESSOR STUDY (NCT00214526), ideally the subject's drug therapy should continue to be consistent with the Global Initiative for Asthma (GINA) Guidelines for the severity of the subject's asthma. Any changes in maintenance levels of asthma medications should be documented.

The goal of this follow-up study is to enroll all subjects who participated in the PREDECESSOR STUDY (NCT00214526). Inclusion of subjects from the treatment arm will allow for the assessment of long-term safety of the Alair procedure for up to 5 years post treatment with the Alair System. Inclusion of subjects from the Control arm will allow for appropriate analysis of long-term effectiveness data for up to 3 years post "treatment".

ELIGIBILITY:
Inclusion Criteria:

1. Subject who participated in the PREDECESSOR STUDY entitled "Multicenter Randomized Clinical Trial of the Alair System for the Bronchial Thermoplasty Treatment of Asthma"(Protocol # 0602-20, NCT00214526).
2. Subject who is able to read, understand, and provide written Informed Consent.
3. Subject who is able to comply with the study protocol, including requirements for taking and abstaining from medications, and complete all study required visits.

Exclusion Criteria:

1. Subject participating in another clinical trial involving respiratory intervention that could affect the outcome measures of this study, either within 6 weeks of study enrollment, or during the study period.
2. Subject with a newly diagnosed (since exiting from the PREDECESSOR STUDY) psychiatric disorder which in the judgment of the investigator could interfere with provision of informed consent, completion of tests, therapy, or follow-up.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2005-03; Primary Completion 2009-12 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Narinder S Shargill, PhD, Study Director — Asthmatx, Inc.
Locations (5):
- Irmandade Santa Casa de Misericordia de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil
- Canada (2):
  - St. Joseph's Healthcare, Hamilton, Ontario
  - Hopital Laval, Laval University, Sainte-Foy, Quebec
- United Kingdom (2):
  - Gartnavel General Hospital, Univ. Glasgow, Glasgow, Scotland
  - Northwest Lung Research Center, Univ. Manchester, Manchester

REFERENCES:
- [Result] Thomson NC, Rubin AS, Niven RM, Corris PA, Siersted HC, Olivenstein R, Pavord ID, McCormack D, Laviolette M, Shargill NS, Cox G; AIR Trial Study Group. Long-term (5 year) safety of bronchial thermoplasty: Asthma Intervention Research (AIR) trial. BMC Pulm Med. 2011 Feb 11;11:8. doi: 10.1186/1471-2466-11-8. PMID 21314924

RESULTS

PARTICIPANT FLOW:
Groups:
- Alair: Alair-treated subjects from AIR PREDECESSOR STUDY (NCT00214526).
- Control: Control subjects from AIR PREDECESSOR STUDY (NCT00214526).
Period: Year 1
Arm/Group | Alair | Control
Started | 45 | 24
Completed | 45 | 24
Not Completed | 0 | 0
Period: Year 2
Arm/Group | Alair | Control
Started | 45 | 24
Completed | 41 | 23
Not Completed | 4 | 1
Not completed — Missed visit but remained in study | 4 | 1
Period: Year 3
Arm/Group | Alair | Control
Started | 45 | 24
Completed | 41 | 21
Not Completed | 4 | 3
Not completed — Withdrawal by Subject | 1 | 3
Not completed — Lost to Follow-up | 1 | 0
Not completed — Missed visit but remained in study | 2 | 0
Period: Year 4
Arm/Group | Alair | Control
Started | 43 | 0 (Control group subjects exited from study after completing Year 3 evaluation.)
Completed | 43 | 0 (Control group subjects exited from study after completing Year 3 evaluation.)
Not Completed | 0 | 0
Period: Year 5
Arm/Group | Alair | Control
Started | 43 | 0 (Control group subjects exited from study after completing Year 3 evaluation.)
Completed | 42 | 0 (Control group subjects exited from study after completing Year 3 evaluation.)
Not Completed | 1 | 0
Not completed — Missed visit but remained in study | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Alair Treatment: Alair treated subjects from PREDECESSOR STUDY (NCT00214526).
  Bronchial Thermoplasty with the Alair System: Treatment of airways with the Alair System in the PREDECESSOR STUDY.
- Total: Total of all reporting groups
Arm/Group | Alair Treatment | Control | Total
Number analyzed (Participants) | 45 | 24 | 69
Age, Continuous [Mean (Standard Deviation); unit: years] | 40 (11.21) | 40.88 (12.13) | 40.30 (11.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 15 | 41
  Male | 19 | 9 | 28
Race/Ethnicity, Customized [Number; unit: participants]
  White | 41 | 22 | 63
  Black | 3 | 2 | 5
  Hispanic | 0 | 0 | 0
  Asian | 1 | 0 | 1
Height (cm) [Mean (Standard Deviation); unit: cm] | 166.17 (9.64) | 164.83 (7.72) | 165.70 (8.99)
Weight (kg) [Mean (Standard Deviation); unit: kg] | 76.37 (23.31) | 77.71 (16.95) | 76.84 (21.20)
Inhaled Corticosteroid Dose [Mean (Standard Deviation); unit: mcg (micrograms)] — Dose of Beclomethasone. All other inhaled corticosteroid doses were converted to their equivalent doses of Beclomethasone.
  mcg (micrograms) | 1291.11 (862.10) | 1135.42 (1030.46) | 1236.96 (919.58)
Long-acting Beta Agonists (LABA) Dose [Mean (Standard Deviation); unit: mcg (micrograms)] — Dose of Salmeterol. All other LABA doses were converted to their equivalent doses of Salmeterol.
  mcg (micrograms) | 108.89 (33.78) | 100.00 (14.74) | 105.80 (28.81)
Methacholine PC20 [Geometric Mean (Full Range); unit: mg/ml] — PC20 is the provocative concentration required to achieve a 20% fall in forced expired volume in one second (FEV1).
  mg/ml | 0.25 [0.2 to 0.4] | 0.28 [0.1 to 0.6] | 0.26 [0.1 to 0.6]
Asthma Control Questionnaire (ACQ) Overall Score [Mean (Standard Deviation); unit: Scores on a scale] — The ACQ has 7 questions (the top scoring 5 symptoms, FEV1% predicted and daily rescue bronchodilator use). Patients are asked to recall how their asthma has been during the previous week and to respond to the symptom and bronchodilator use questions on a 7-point scale (0=no impairment, 6= maximum impairment). Clinic staff score the FEV1% predicted on a 7-point scale. The questions are equally weighted and the ACQ score is the mean of the 7 questions and therefore between 0 (totally controlled) and 6 (severely uncontrolled).
  Scores on a scale
    LABA Stable | 1.39 (0.68) | 1.29 (0.7) | 1.36 (0.89)
    LABA Withdrawal | 2.50 (0.97) | 2.08 (0.90) | 2.35 (0.96)
Asthma Quality of Life Questionnaire (AQLQ) Score [Mean (Standard Deviation); unit: Scores on a scale] — There are 32 questions in the AQLQ and they are in 4 domains (symptoms, activity limitation, emotional function and environmental stimuli). Patients are asked to think about how they have been during the previous two weeks and to respond to each of the 32 questions on a 7-point scale (7 = not impaired at all - 1 = severely impaired). The overall AQLQ score is the mean of all 32 responses and the individual domain scores are the means of the items in those domains.
  Scores on a scale
    LABA Stable | 5.65 (0.99) | 5.62 (0.92) | 5.64 (0.96)
    LABA Withdrawal | 4.88 (1.30) | 4.84 (1.40) | 4.86 (1.33)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Any Respiratory Adverse Event
Description: There is not one specific primary outcome measure. The primary objective of this study is to gather additional, longer-term safety data in subjects who participated in the AIR Trial (Protocol #0602-20), called the AIR PREDECESSOR STUDY in the AIR Extension Report (NCT00214526). The 'Percentage of Subjects with any Respiratory Adverse Event' was chosen to be the primary outcome measure because it is the first described in the final study report.
Time Frame: 12 Month periods out to 5 years
Measure: Count of Participants; unit: Participants
Groups:
- Alair Year 1: Alair treated subjects from PREDECESSOR STUDY (NCT00214526), Year 1.
  Bronchial Thermoplasty with the Alair System: Treatment of airways with the Alair System in the PREDECESSOR STUDY
- Alair Year 2: Alair treated subjects from PREDECESSOR STUDY (NCT00214526), Year 2.
  Bronchial Thermoplasty with the Alair System: Treatment of airways with the Alair System in the PREDECESSOR STUDY
- Alair Year 3: Alair treated subjects from PREDECESSOR STUDY (NCT00214526), Year 3.
  Bronchial Thermoplasty with the Alair System: Treatment of airways with the Alair System in the PREDECESSOR STUDY
- Alair Year 4: Alair treated subjects from PREDECESSOR STUDY (NCT00214526), Year 4.
  Bronchial Thermoplasty with the Alair System: Treatment of airways with the Alair System in the PREDECESSOR STUDY
- Alair Year 5: Alair treated subjects from PREDECESSOR STUDY (NCT00214526), Year 5.
  Bronchial Thermoplasty with the Alair System: Treatment of airways with the Alair System in the PREDECESSOR STUDY
- Control Year 1: Control group subjects from PREDECESSOR STUDY (NCT00214526) Year 1.
- Control Year 2: Control group subjects from PREDECESSOR STUDY (NCT00214526) Year 2.
- Control Year 3: Control group subjects from PREDECESSOR STUDY (NCT00214526) Year 3.
Arm/Group | Alair Year 1 | Alair Year 2 | Alair Year 3 | Alair Year 4 | Alair Year 5 | Control Year 1 | Control Year 2 | Control Year 3
Number analyzed (Participants) | 45 | 45 | 43 | 43 | 42 | 24 | 24 | 21
Participants | 38 | 24 | 24 | 23 | 22 | 18 | 13 | 12

2. Other Pre Specified Outcome: Health Care Usage
Time Frame: 12 Month periods out to 5 years
Measure: Mean (Standard Deviation); unit: Number events per subject
Arm/Group | Alair Year 1 | Alair Year 2 | Alair Year 3 | Alair Year 4 | Alair Year 5 | Control Year 1 | Control Year 2 | Control Year 3
Number analyzed (Participants) | 45 | 45 | 43 | 43 | 42 | 24 | 24 | 21
Number events per subject
  Hospitalizations for Respiratory Symptoms | 0.07 (0.25) | 0.07 (0.25) | 0.07 (0.46) | 0.02 (0.15) | 0.02 (0.15) | 0.00 (0.00) | 0.00 (0.00) | 0.05 (0.22)
  Emergency Room (ER) Visits for Respiratory Symptoms | 0.04 (0.21) | 0.07 (0.25) | 0.07 (0.34) | 0.14 (0.47) | 0.05 (0.22) | 0.00 (0.00) | 0.13 (0.34) | 0.14 (0.85)
  Unscheduled Physician Office Visits for Respiratory Symptoms | 0.42 (0.72) | 0.18 (0.44) | 0.44 (0.70) | 0.70 (1.21) | 0.48 (0.94) | 0.42 (0.72) | 0.25 (0.74) | 0.29 (0.64)

3. Other Pre Specified Outcome: Number of Respiratory Adverse Events
Description: Number of respiratory adverse events per subject
Time Frame: 12 Month periods out to 5 years
Measure: Mean (Standard Deviation); unit: Number events per subject
Arm/Group | Alair Year 1 | Alair Year 2 | Alair Year 3 | Alair Year 4 | Alair Year 5 | Control Year 1 | Control Year 2 | Control Year 3
Number analyzed (Participants) | 45 | 45 | 43 | 43 | 42 | 24 | 24 | 21
Number events per subject | 4.5 (4.2) | 1.2 (1.6) | 1.3 (1.9) | 1.2 (1.6) | 1.1 (2.2) | 3.1 (3.7) | 1.2 (1.1) | 1.3 (1.6)

4. Other Pre Specified Outcome: Forced Expiratory Volume in 1 Second (FEV1) - % Predicted
Time Frame: 12 Month periods out to 5 years
Measure: Mean (Standard Deviation); unit: percentage predicted
Arm/Group | Alair Year 1 | Alair Year 2 | Alair Year 3 | Alair Year 4 | Alair Year 5 | Control Year 1 | Control Year 2 | Control Year 3
Number analyzed (Participants) | 40 | 37 | 35 | 36 | 35 | 19 | 23 | 21
percentage predicted
  Pre-Bronchodilator Off-LABA | 76.0 (14.0) | 73.5 (15.0) | 73.9 (12.6) | 74.3 (15.0) | 70.6 (14.6) | 71.6 (11.6) | 74.8 (10.6) | 70.1 (16.9)
  Post-Bronchodilator Off-LABA | 84.5 (13.3) | 85.0 (13.1) | 85.1 (11.6) | 84.6 (14.2) | 83.5 (13.5) | 82.2 (8.5) | 86.3 (9.7) | 80.7 (19.8)

ADVERSE EVENTS:
Time Frame: Year 1 Post-Treatment out to 5 years for Alair participants, Year 1 Post-Treatment out to 3 years for Control participants.
Groups:
- Alair - Year 1; Alair - Year 2; Alair - Year 3; Alair - Year 4; Alair - Year 5: Alair treated subjects from PREDECESSOR STUDY (NCT00214526).
- Control - Year 1; Control - Year 2; Control - Year 3: Control treated subjects from PREDECESSOR STUDY (NCT00214526).
Arm/Group | Alair - Year 1 | Alair - Year 2 | Alair - Year 3 | Alair - Year 4 | Alair - Year 5 | Control - Year 1 | Control - Year 2 | Control - Year 3
All-Cause Mortality (participants affected / at risk) | 0/45 | 0/45 | 0/43 | 0/43 | 0/42 | 0/24 | 0/23 | 0/21
Serious Adverse Events (participants affected / at risk) | 4/45 | 4/45 | 3/43 | 3/43 | 3/42 | 2/24 | 0/23 | 1/21
Other Adverse Events (participants affected / at risk) | 42/45 | 23/45 | 23/43 | 22/43 | 22/42 | 19/24 | 12/23 | 11/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alair - Year 1 (N=45) | Alair - Year 2 (N=45) | Alair - Year 3 (N=43) | Alair - Year 4 (N=43) | Alair - Year 5 (N=42) | Control - Year 1 (N=24) | Control - Year 2 (N=23) | Control - Year 3 (N=21)
Left Leg Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Non-respiratory
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Respiratory
Lower Respiratory Tract Infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Respiratory
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Respiratory
Knee surgery (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Non-respiratory
Nasosinusal polyps (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Respiratory
Lung infection pseudomonal (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Respiratory
Diverticulitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Non-respiratory
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Non-respiratory
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Non-respiratory
Tubal obstruction (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Non-respiratory
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Non-respiratory
Sepsis (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Non-respiratory
Headache (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Non-respiratory
Chest discomfort (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) — Respiratory
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Respiratory
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) — Respiratory
Respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Respiratory
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Respiratory
Calculus urinary (Renal and urinary disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Non-respiratory
Laparotomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Non-respiratory
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alair - Year 1 (N=45) | Alair - Year 2 (N=45) | Alair - Year 3 (N=43) | Alair - Year 4 (N=43) | Alair - Year 5 (N=42) | Control - Year 1 (N=24) | Control - Year 2 (N=23) | Control - Year 3 (N=21)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Non-Respiratory
Nausea (Gastrointestinal disorders) | 4 (4) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Non-Respiratory
Ear infection (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Non-Respiratory
Influenza (Infections and infestations) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0) — Non-Respiratory
Sinusitis (Infections and infestations) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) — Non-Respiratory
Tonsillitis (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Non-Respiratory
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (3) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Non-Respiratory
Headache (Nervous system disorders) | 13 (36) | 1 (1) | 1 (1) | 2 (2) | 1 (2) | 4 (4) | 0 (0) | 0 (0) — Non-Respiratory
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (5) | 7 (8) | 7 (8) | 6 (8) | 0 (0) | 2 (2) | 1 (4) — Respiratory
Chest discomfort (Respiratory, thoracic and mediastinal disorders) | 7 (9) | 2 (2) | 3 (4) | 1 (1) | 2 (2) | 3 (5) | 1 (2) | 1 (1) — Respiratory
Cough (Respiratory, thoracic and mediastinal disorders) | 17 (29) | 4 (5) | 2 (2) | 3 (4) | 2 (6) | 8 (9) | 0 (0) | 3 (3) — Respiratory
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 20 (40) | 4 (4) | 4 (4) | 4 (5) | 4 (7) | 12 (22) | 2 (2) | 3 (3) — Respiratory
Lower respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 2 (3) | 0 (0) | 3 (3) | 1 (1) — Respiratory
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 13 (21) | 2 (2) | 0 (0) | 0 (0) | 1 (2) | 5 (6) | 0 (0) | 0 (0) — Respiratory
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Respiratory
Nocturnal dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) — Respiratory
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) — Respiratory
Productive cough (Respiratory, thoracic and mediastinal disorders) | 9 (14) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 6 (6) | 0 (0) | 0 (0) — Respiratory
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) — Respiratory
Respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 3 (3) | 5 (6) | 3 (6) | 2 (3) | 5 (6) | 2 (4) | 1 (1) — Respiratory
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) — Respiratory
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (3) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 0 (0) — Respiratory
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Respiratory
Tracheobronchitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (3) — Respiratory
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 10 (15) | 11 (17) | 8 (13) | 8 (13) | 4 (5) | 2 (3) | 3 (5) | 4 (7) — Respiratory
Wheezing (Respiratory, thoracic and mediastinal disorders) | 14 (19) | 2 (3) | 3 (5) | 3 (4) | 2 (2) | 4 (6) | 1 (1) | 1 (1) — Respiratory

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less